CLINICAL TRIAL: NCT03636191
Title: The Effect of Lactobacillus Rhamnosus (LGG®) on the Defence Against Pathogens in the Upper Respiratory Tract in Healthy Children - a Single-center, Randomized, Double-blind, Placebo-controlled Study With 16 Weeks Intervention.
Brief Title: The Effect of a Probiotic on Upper Respiratory Tract Infections
Acronym: PIP-U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: Onorach Clinical (Unknown); CPS Research (Unknown)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-IM-030
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Infections, Upper Respiratory Tract
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic strain
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic strain — Lactobacillus
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, two-armed, parallel-group study in healthy children aged 2-6 years. The study will investigate the effect of daily intake of a probiotic on Upper Respiratory Tract Infections (URTI) during a 16-week intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2-6 years, both inclusive, at the time of informed consent
2. No URTI at the time of inclusion as assessed by a GP
3. Attending day-care with at least 10 children or primary school with at least 10 children in the class for at least 20 hours a week
4. Generally healthy as determined by a GP
5. Guardian consents to participate in the study and to comply with all its procedures

Exclusion Criteria:

1. Any known concomitant chronic infections, chronic systemic diseases, autoimmune diseases (e.g. asthma), immunodeficiency, metabolic diseases, chronic respiratory tract diseases including respiratory allergies and cystic fibrosis, congenital cardiac defects.
2. Suspected or challenge-proved food allergy
3. Use of any prescribed immune suppressive medications at enrolment
4. Use of oral or IV antibiotics in the 1 month before randomisation
5. Not willing to exclude pre/pro/synbiotics during the study
6. Intake of Echinacea, high dose vitamins or Zinc four weeks before and during the study period.
7. Language limitations regarding interviews or questionnaires
8. Participation in other clinical studies in the last 2 months
9. Planning extensive travel (for >1 month) during the duration of the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 619 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
The incidence of URTI | 16 weeks
  The incidence of URTI measured as the number of URTI episodes diagnosed by a GP according to the prespecified, well-defined criteria, adjusted for sample size.

SECONDARY OUTCOMES:
The incidence of URTI with pathogens | 16 weeks
  The incidence of URTI measured as the number of URTI episodes diagnosed by a GP according to the prespecified, well-defined criteria, for which a pathogen is identified in nasal swabs, adjusted for sample size.
The Number of days with URTI symptoms | 16 weeks
  The number of days with URTI symptoms for URTIs that were diagnosed by a GP, adjusted for sample size.
The number of days with temperature ≥ 38 °C | 16 weeks
  The number of days with temperature ≥ 38 °C during an URTI episode, which was diagnosed by a GP, adjusted for sample size.
WURSS-K score | 16 weeks
  The Area under Curve for daily Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K) score (range: not sick - very sick) during an URTI episode, which was diagnosed by a GP, adjusted for sample size.
The number of subjects with one or more episode of URTI | 16 weeks
  The number of subjects with one or more episode of URTI, which was diagnosed by a GP, adjusted for sample size.
The number of days of absence from daycare or primary school | 16 weeks
  The number of days of absence from daycare or primary school during an URTI, which was diagnosed by a GP, adjusted for sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Crawford, DRCOG, Principal Investigator — CPS Research
Locations (1):
- CPS Research, Glasgow, United Kingdom

REFERENCES:
- [Derived] Damholt A, Keller MK, Baranowski K, Brown B, Wichmann A, Melsaether C, Eskesen D, Westphal V, Arltoft D, Habicht A, Gao Q, Crawford G. Lacticaseibacillus rhamnosus GG DSM 33156 effects on pathogen defence in the upper respiratory tract: a randomised, double-blind, placebo-controlled paediatric trial. Benef Microbes. 2022 Feb 28;13(1):13-23. doi: 10.3920/BM2021.0065. Epub 2021 Dec 13. PMID 34895109